CLINICAL TRIAL: NCT05494346
Title: Prospective Multicenter Clinical Investigation Evaluating the Performance and Safety of Gilbert Laboratories' Decongestant Seawater Spray Pocket Valve Enriched With Essential Oils
Brief Title: Safety and Performance Assessment of the Decongestant Seawater Spray Pocket Valve Enriched With Essential Oils in Patients With Acute Rhinitis Associated With Nasal Obstruction: "DEVALPO"
Acronym: DEVALPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Gilbert (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A01898-33
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Acute Rhinitis; Nasal Obstruction; Rhinosinusitis; Rhinopharyngitis; Allergic Rhinitis
MeSH Terms: conditions — Common Cold; Nasal Obstruction; Rhinosinusitis; Nasopharyngitis; Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Patients with peak nasal flow performed (Other): This arm is made up of major patients. Nasal flow point measurements will be performed at D0 and D3.
  Interventions: Device: Measurement of peak nasal flow.
- Arm B: No peak nasal flow (No Intervention): This arm is made up of minor patients. Unlike arm A, nasal flow measurements will not be performed at D0 and D3.

INTERVENTIONS:
Device: Measurement of peak nasal flow. — Peak nasal flow measurements will be performed before and after the first use of the spray at D0, as well as after the use of the spray at the medical office at D3 (only for arm A).
  Arms: Arm A: Patients with peak nasal flow performed

SUMMARY:
The purpose of this pre-market clinical investigation is to assess the safety and the performance of decongestant seawater spray pocket valve enriched with essential oils by Gilbert Laboratories. The study will evaluate the results of acute rhinitis associated with nasal obstruction using the decongestant seawaterspray pocket valve enriched with essential oils over a 8 day period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient ≥ 12 years.
* 2. Patient with acute rhinitis associated with nasal obstruction during infectious episodes such as rhinopharyngitis (cold), rhinosinusitis, or during non-infectious episodes such as allergic rhinitis.
* 3. a. Informed adult patient who has given written consent prior to any study specific procedure. b. Informed minor patient who has given assent and whose legal guardians have given written consent prior to any study-specific procedure.
* 4. Patient able to meet the study requirements for monitoring, spray use, and questionnaire completion.
* 5. Patient affiliated to a social security scheme.

Exclusion Criteria:

* 1. Pregnant and/or breastfeeding woman
* 2. Hypersensitivity to seawater and/or known allergies to any of the ingredients of the spray.
* 3. Diseases causing narrowing of the airways (e.g. asthma, chronic obstructive pulmonary disease (COPD)) and/or respiratory insufficiency.
* 4. Patients with uncontrolled asthma (GINA score greater than or equal to 4)
* 5. Patients undergoing allergy desensitization
* 6. Patients suffering from chronic nasal obstruction due to a deformation of the nasal wall or nasal polyps. creams or gels.
* 7. Patients taking local and systemic vasoconstrictors, corticosteroids, nonsteroidal anti-inflammatory drugs (NSAIDs), antibiotics, and local antiseptics.
* 8. Concomitant use of other nasal sprays, essential oils for local nasal use, creams, or gels for the nose.
* 9. Patients under guardianship, conservatorship, or legal protection.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Performance of the Gilbert Laboratories pocket valve spray. | From Day 0 to Day 3
  Proportion of patient presenting a change of the symptom "nasal obstruction" by at least 1 pt, in the SNOT22 Test (item 22), between Day 0 (at inclusion in the office before use of the spray) and Day 3 (in the evening after last daily use of the spray).
  This item is scaled from 0 to 5, 5 being the worst value.

SECONDARY OUTCOMES:
Change of nasal obstruction between Day 0 and Day 3 | From Day 0 to Day 3
  Proportion of patients with a change in Peak Inspiratory Nasal Flow value of at least 30 L/min between Day 0 (before use of the spray) and Day 3 (after use of the spray) (arm A).
  [0 - 350 L/min] 350 L/min means a better outcome.
Immediate change of nasale obstruction at D0 on first use (Arm A) | At Day 0
  Proportion of patients with a change in Peak Inspiratory Nasal Flow value of at least 30 L/min from pre- to post-spray measurements at Day 0 (arm A).
  [ 0 - 350 L/min] 350 L/min means a better outcome.
Subjective feeling of reduced nasal obstruction on each day of use (arms A+B). | From Day 0 to Day 6
  Proportion of patients with a reduction in the symptom "nasal obstruction" of at least 1pt, on SNOT22 (Sino-Nasal Outcome Test 22), and on each day of use (from Day 0 to Day 6) (arms A+B).
  This item is scaled from 0 to 5, 5 being the worst value.
Subjective feeling of nasal cavity cleansing (freshness) each day of use (arms A+B). | From Day 0 to Day 6
  Proportion of patients who experienced nasal cavity cleansing (feeling of freshness), on Patient Questionnaire, and on each day of use (from Day 0 to Day 6) (arms A+B).
Subjective feeling of nasal secretion thinning on each day of use (arms A+B). | From Day 0 to Day 6
  Proportion of patients with a change in the symptom "thick nasal discharge" of at least 1pt, on SNOT22, and on each day of use (Day 0 to Day 6) (arms A+B).
  This item is scaled from 0 to 5, 5 being the worst value.
Subjective feeling of relief of nasal irritation (mucous membrane) on each day of use (arms A+B). | From Day 0 to Day 6
  Proportion of patients who experienced relief of nasal (mucosal) irritation, on each day of use (Day 0 to Day 6) (arms A+B).
Subjective feeling of relief of nasal itching on each day of use (arms A+B). | From Day 0 to Day 6
  Proportion of patients who experienced relief of nasal itching, on Patient Questionnaire, and on each day of use (Day 0 to Day 6) (arms A+B).
Speed of action at which the patient feels (subjectively) a decrease in nasal obstruction at D0 and D3 (arms A+B). | At Day 0 and Day 3
  Proportion of patients with a change in immediate nasal obstruction after use of the spray, on Patient Questionnaire, at Day 0 and Day 3 (arms A+B).
Speed of action at which the patient feels (subjectively) a purification of his nasal cavities (sensation of freshness) at D0 and D3 (arms A+B). | At Day 0 and Day 3
  Proportion of patients who experienced immediate nasal cleansing (feeling of freshness) after use of the spray at Day 0 and Day 3 (arms A+B).
Improvement in the patient's quality of life after 7 days of use (arms A+B). | From Day 0 to Day 6
  Proportion of patients who experienced an improvement in quality of life, defined as an increase of at least 1pt on a scale of 0-10 between Day 0 and Day 6 (A+B arm).
  10 mean a better value.
Patient satisfaction with the medical device after 7 days of use (arm A+B). | At Day 6
  Proportion of patients satisfied with the medical device, on a 4-point scale, at Day 6 (arm A+B).
  The better value is "very satisfied" and the worst value is "very unsatisfied". Proportion of patients who would recommend the medical device at Day 6 (arms A+B).
  Proportion of patients who will continue to use the medical device , and the reason if not, (arms A+B).
Facility of use of the medical device after 7 days of use (arm A+B) | At Day 6
  Proportion of patients who find the medical device easy to use, on day 6 (Arms A+B)
Evolution of the overall severity of symptoms (arm A+B). | At Day 0 and Day 3
  Mean SNOT22 score on each day. Comparison of SNOT22 score at Day 3 versus Day 0 baseline (arms A+B).
  [ 0 to 220 ] 0 is the better value.
Sensations of tingling and transient irritation (arms A+B). | From Day 0 to Day 6
  Proportion of patients with at least 1 adverse event between 1st and last use of the medical device among the following adverse events (arms A+B):
  * Tingling sensations
  * Sensations of transient irritation
All adverse events reported by patients using the pocket valve spray after 7 days of use (arm A+B). | From Day 0 to Day 7
  All adverse events reported by the patient during the study (arm A+B).

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Cabinet Médical, Blainville-sur-Orne
  - Cabinet Médical Caen, Caen
  - MSP du Haut Anjou, Châteauneuf-sur-Sarthe
  - Cabinet Médical Gainneville, Gainneville
  - ALYATEC, Strasbourg

IPD SHARING:
Plan to Share IPD: No